CLINICAL TRIAL: NCT00025662
Title: Ex Vivo Selective Depletion of Alloreactive Donor T-Lymphocytes Using "RFT5-SMPT-dgA": Reducing GVHD Risk Associated With Matched, Nonmyeloablative, Stem Cell Transplant for Hematologic Malignancies in Older Adults
Brief Title: Selective T-Cell Depletion to Reduce GVHD (Patients) Receiving Stem Cell Tx to Treat Leukemia, Lymphoma or MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010162; 01-H-0162 (Other: NIH); NCT00016484 (obsolete NCT alias)
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-09

CONDITIONS: Graft vs Host Disease; Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid; Leukemia, Myelomonocytic, Chronic; Leukemia, Lymphocytic; Lymphoma; Lymphoma, Mantle-cell; Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: Peripheral Blood Stem Cell; Melphalan; Fludarabine; Donor Apheresis; Non-Myeloablative; MDS; Chronic Myeloid Leukemia; CML; Chronic Lymphocytic Leukemia; CLL; Lymphoma; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Mantle Cell Lymphoma; Acute Myelogenous Leukemia (AML); Chronic Myeloid Leukemia (CML); Chronic Lymphocytic Leukemia (CLL); Myelodysplasia (MDS); Acute Lymphoblastic Leukemia (ALL); Bone Marrow Transplant
MeSH Terms: conditions — Graft vs Host Disease; Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid; Leukemia, Myelomonocytic, Chronic; Leukemia, Lymphoid; Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — RFT5-SMPT-dgA immunotoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RFT5-SMPT-dgA Isolex system (Experimental): RFT5-SMPT-dgA, a specific anti-interleukin-2 receptor immunotoxin used in allogeneic stem cell transplantation (SCT) in older patients with hematologic malignancies using a graft manipulation process
  Interventions: Drug: RFT5-SMPT-dgA; Drug: Isolex system

INTERVENTIONS:
Drug: RFT5-SMPT-dgA — A specific anti-interleukin-2 receptor immunotoxin
  Other Names: anti-interleukin-2 receptor immunotoxin
Drug: Isolex system — CD34 selection/ T cell depletion used this system
  Other Names: Nexell Isolex system

SUMMARY:
This study will evaluate the safety and effectiveness of stem cell transplantation in which the donors T lymphocytes have undergone "selective depletion." Certain patients with cancers of the blood undergo transplantation of donated stem cells to generate new and normally functioning bone marrow. In addition to producing the new bone marrow, the donor's T-lymphocytes also fight any tumor cells that might have remained in the body. This attack on tumor cells is called a "graft-versus-leukemia" (GVL) effect. However, another type of T-lymphocyte from the donor may cause what is called "graft-versus-host-disease" (GVHD), in which the donor cells recognize the patient's cells as foreign and mount an immune response to reject them. Selective depletion is a technique that was developed to remove the T-lymphocytes that cause harmful GVHD, while keeping those that produce the desirable GVL effect.

DETAILED DESCRIPTION:
Despite improved prophylaxis and treatment, graft-versus-host disease (GVHD) remains a major complication after allogeneic stem cell transplantation. Although the most effective way to prevent GVHD is T cell depletion, this process results in poor immune function leading to increased rates of relapse, graft rejection, and post-transplant infections. Ideally, a method of removing GVHD- producing effector cells while retaining a broad T cell repertoire, including preservation of 3rd party, antiviral and anti-tumor responses would be desirable. Preclinical studies from our lab have demonstrated that alloreactive T cells can be selectively removed from the donor lymphocyte pool in vitro with the use of a specific immunotoxin directed against the interleukin-2 receptor.

To test this clinically, we will perform nonmyeloablative allogeneic stem cell transplants in older patients with hematologic malignancies. Although these patients can be cured with this approach, they have significant morbidity and mortality from GVHD. At our institution, nonmyeloablative transplantation is associated with an incidence of grade II-IV acute GVHD of approximately 50%. Although well tolerated in younger patients, patients over the age of 50 years have a transplant-related mortality (TRM) of approximately 35%, which is mostly related to GVHD. Through selective depletion of alloreactive donor lymphocytes, we hope to reduce GVHD mortality, while preserving the transplant efficacy.

Patients receive a reduced intensity preparative regimen, followed by a mobilized peripheral blood stem cell allograft from an HLA-identical sibling donor, containing "selectively-depleted" donor lymphocytes. To obtain such a graft, colony stimulating factor (G-CSF)-mobilized peripheral blood from the donor undergoes a positive cluster of differentiation (CD34) selection followed by a negative T cell selection using the "Nexell" Isolex 300i system. This stem cell-rich, T cell-depleted product will contain a CD34+ cell dose of at least 5x10(6)/kg. The unabsorbed fraction, remaining after the positive CD34 selection, is then co-cultured for 72 hours with irradiated lymphocytes from the patient. The immunotoxin, RFT5-SMPT-dgA, is added during the last 24 hours of culture to remove alloreacting cells. The washed T cell product (CD3+ cell dose of 1-4 x 10(8)/kg) is cryopreserved. Following the preparative regimen, the patient receives successive infusions of the stem cell product and selected lymphocytes. All patients receive standard post transplant immunosuppression with cyclosporine for a minimum of 30 days, followed by dose reduction depending on the degree of donor lymphocyte chimerism.

The primary end point of this study is the incidence and severity of acute GVHD. We will also examine the incidence of chronic GVHD, engraftment, degree of donor-host chimerism, transplant related morbidity and mortality, as well as disease-free and overall survival. Stopping rules will minimize the risk of untoward or unexpected side effects.

ELIGIBILITY:
- INCLUSION CRITERIA: PATIENT

* Ages 50-75 years
* Relapsed CML in chronic or accelerated phase after therapy with STI-571 (Gleevec)
* Acute lymphoblastic leukemia (ALL), all patients in complete or partial remission. Exceptions: T cell ALL
* Acute myelogenous leukemia (AML): AML in first complete or partial remission including AML secondary to chemotherapy or prior hematological disease such as myelodysplastic syndrome, and myeloproliferative disorder.
* Myelodysplastic syndromes: (1) refractory anemia with excess of blasts (RAEB), (2) refractory anemia with excess blasts in transformation (RAEBT), (3) MDS with poor risk cytogenetics defined by a complex karyotype (greater than or equal to three anomalies) or chromosome 7 abnormalities, (4) secondary MDS after prior cytotoxic or radiation therapy, or (5) chronic myelomonocytic leukemia (CMML)
* Chronic lymphocytic leukemia (CLL) and prolymphocytic leukemia, refractory to nucleoside analog therapy, with either progressive bulky disease or anemia (less than 10 g/dl) or thrombocytopenia (less than 100,000/microliter) not due to recent chemotherapy
* Mantle cell lymphoma
* Relapsed intermediate- or high-grade non-Hodgkin's lymphoma: (1) post autologous marrow or PBSC transplant, or (2) chemorefractory relapse. Exceptions: T cell NHL
* Relapse Hodgkin's disease: (1) post autologous marrow or PBSC transplant, or (2) chemorefractory relapse
* Low-grade follicular or small lymphocytic lymphoma: (1) relapsed following conventional chemotherapy, (2) relapsed following autologous marrow or PBSC transplant, or (3) chemoresistant disease
* Life expectancy greater than 3 months
* Ability to comprehend the investigational nature of the study and provide informed consent
* Availability of an HLA-identical family donor, 18 to 75 years old
* INCLUSION CRITERIA:

DONOR

* HLA identical family donor, 18 to 75 years old
* Fit to receive G-CSF and give peripheral blood stem cells (normal blood count, normotensive, no history of stroke, no history of severe heart disease)
* Ability to comprehend the investigational nature of the study and provide informed consent
* EXCLUSION CRITERIA:

RECIPIENT

* Pregnant or lactating
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or more
* Major anticipated illness or organ failure incompatible with survival from PBSC transplant
* Diffusion Capacity fir carbon monoxide (DLCO) less than 60% predicted
* Left ventricular ejection fraction less than 40%, or any angina.
* Absolute lymphocyte count less than 300/mm(3)
* Serum creatinine greater than 2.5 mg/dl
* Serum bilirubin greater than 4 mg/dl, transaminases greater than 5x upper limit of normal
* HIV positive
* Other malignant diseases liable to relapse or progress within 2 years
* EXCLUSION CRITERIA:

DONOR

* Pregnant or lactating
* HIV positive. Donors who are positive for Hepatitis B Virus, Hepatitis C Virus or human t-cell lymphoma virus (HTLV) will be used at the discretion of the investigator and with appropriate consent of the recipient
* Donor unfit to receive G-CSF and undergo apheresis (uncontrolled hypertension, history of heart failure or unstable angina, platelet count less than 90,000/cu mm)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-05; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A. J Barrett, MD, Study Chair — NHLBI, NIH
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barrett J, Solomon S. The transition from bench to bedside: lessons learned in the creation of a new T-cell product for the clinic. Cytotherapy. 2004;6(6):593-5. doi: 10.1080/14653240410011936. PMID 15764025
- [Background] Solomon SR, Tran T, Carter CS, Donnelly S, Hensel N, Schindler J, Bahceci E, Ghetie V, Michalek J, Mavroudis D, Read EJ, Vitetta ES, Barrett AJ. Optimized clinical-scale culture conditions for ex vivo selective depletion of host-reactive donor lymphocytes: a strategy for GvHD prophylaxis in allogeneic PBSC transplantation. Cytotherapy. 2002;4(5):395-406. doi: 10.1080/146532402320775982. PMID 12473206
- [Background] Mielke S, Solomon SR, Barrett AJ. Selective depletion strategies in allogeneic stem cell transplantation. Cytotherapy. 2005;7(2):109-15. doi: 10.1080/14653240510018172. PMID 16040390
- [Result] Solomon SR, Mielke S, Savani BN, Montero A, Wisch L, Childs R, Hensel N, Schindler J, Ghetie V, Leitman SF, Mai T, Carter CS, Kurlander R, Read EJ, Vitetta ES, Barrett AJ. Selective depletion of alloreactive donor lymphocytes: a novel method to reduce the severity of graft-versus-host disease in older patients undergoing matched sibling donor stem cell transplantation. Blood. 2005 Aug 1;106(3):1123-9. doi: 10.1182/blood-2005-01-0393. Epub 2005 Apr 7. PMID 15817673
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2001-H-0162.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 9/21/01 to 11/14/05 Location: Quaternary referral institute
Pre-assignment Details: 2 enrolled patients were not transplanted: one, because of donor refusal and the other because she was transplanted elsewhere
Groups:
- "RFT5-SMPT-dgA", an Anti-interleukin, Used in Transplants: Ex vivo selective depletion of alloreactive donor T lymphocytes utilizing "RFT5-SMPT-dgA", a specific anti-interleukin-2 receptor immunotoxin in matched, nonmyeloablative, peripheral blood stem cell transplantation for hematologic malignancies in older adults
Period: Overall Study
Arm/Group | "RFT5-SMPT-dgA", an Anti-interleukin, Used in Transplants
Started | 25
Completed | 22 (One patient who received a transplant did not meet eligibility and was a special exemption.)
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Technical failure of manipulation | 1

BASELINE CHARACTERISTICS:
Groups:
- RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants: Ex vivo selective depletion of alloreactive donor T lymphocytes utilizing RFT5-SMPT-dgA, a specific anti-interleukin-2 receptor immunotoxin in HLA-matched, nonmyeloablative, peripheral blood stem cell transplantation for hematologic malignancies in older adults
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 22

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality
Description: Nonrelapse mortality in the first 100 days of transplant expressed as a percentage of the total subjects.
  This is different from outcome measure 3 (Cumulative Nonrelapse Mortality), which is cumulative non relapse mortality till December 2011.
Time Frame: 100 days after stem cell infusion
Population: all 22 patients who received a selectively depleted allogeneic transplant, including one who was a special exemption for not meeting full eligibility criteria
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
percentage of participants | 4.5 [0 to 13.25]

2. Secondary Outcome: Overall Survival
Description: Percent overall survival (actuarial) at analysis in Dec 2011.
Time Frame: Dec 2011.
Population: all patients who received the selectively depleted transplant including one special exemption
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
percentage of participants | 4.5 [0 to 13.3]

3. Secondary Outcome: Cumulative Non Relapse Mortality
Description: Percent non relapse mortality (actuarial) at analysis in Dec 2011
Time Frame: Dec 2011.
Population: All patients who received the selectively depleted transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
percentage of participants | 40.9 [20.4 to 61.5]

4. Other Pre Specified Outcome: Acute GVHD (Any Grade) Using the CIBMTR Grading System.
Description: Proportion of patients with acute GVHD, grade 1 to 4
Time Frame: 100 days from transplant
Population: All 22 subjects who received the selectively depleted transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
percentage of participants | 54.5 [33.7 to 75.4]

5. Other Pre Specified Outcome: Acute GVHD (Grade 3 or 4) Using the CIBMTR Grading System.
Time Frame: 100 days from transplant
Population: All 22 patients who received the selectively depleted transplant
Measure: Number; unit: percentage of participants
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Number analyzed (Participants) | 22
percentage of participants | 18.2

ADVERSE EVENTS:
Time Frame: The adverse event reporting was collected for 7 years.
Arm/Group | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants
Serious Adverse Events (participants affected / at risk) | 22/22
Other Adverse Events (participants affected / at risk) | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | RFT5-SMPT-dgA, an Anti-interleukin, Used in Transplants (N=22)
Non relapse deaths (Immune system disorders) | 8/8 (8)
Relapse deaths (Immune system disorders) | 10/10 (10)
Hospitalization (Immune system disorders) | 4/4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes